CLINICAL TRIAL: NCT01182090
Title: OPEN SURGERY VS LAPAROSCOPY IN SURGERY OF PELVIC ORGAN PROLAPSE
Brief Title: Surgical Correction of Pelvic Organ Prolapse
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Luigi Mearini, senior assistant, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPerugia
Record Dates: First submitted 2010-08-12; First posted 2010-08-16 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2010-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; colposacropexy; surgery
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolapse repair by open approach (Active Comparator): Correction of urogenital prolapse by open surgery approach
  Interventions: Procedure: Colposacropexy
- Prolapse repair by laparoscopic approach (Active Comparator): Correction of urogenital prolapse by laparoscopic approach
  Interventions: Procedure: Colposacropexy

INTERVENTIONS:
Procedure: Colposacropexy — In open approach the anterior vaginal wall is dissected from the bladder to expose a vaginal wall area of at least 3 x 5 cms where the mesh will be attached with four-five Polyglycolic 0 sutures. The procedure is repeated for the posterior vaginal wall, where the mesh will be attached with three-four Polyglycolic 0 sutures. The sacral promontory surface is prepared and 1 or 2 non-reabsorbable 0.0 sutures are placed into the sacral periosteum about 2 cm below the promontory. A sub-peritoneal tunnel is created through which meshes are passed avoiding traction to the sacrum. The peritoneum is closed over the meshes.
  Arms: Prolapse repair by open approach
Procedure: Colposacropexy — In laparoscopic approach the anterior vaginal wall is dissected from the bladder to expose a vaginal wall area of at least 3 x 5 cms where the mesh will be attached with four-five Polyglycolic 0 sutures. The procedure is repeated for the posterior vaginal wall, where the mesh will be attached with three-four Polyglycolic 0 sutures. The sacral promontory surface is prepared and 1 or 2 non-reabsorbable 0.0 sutures are placed into the sacral periosteum about 2 cm below the promontory. A sub-peritoneal tunnel is created through which meshes are passed avoiding traction to the sacrum. The peritoneum is closed over the meshes.
  Arms: Prolapse repair by laparoscopic approach

SUMMARY:
Objective:

This prospective randomized trial evaluated outcomes of colposacropexy performed either by open or by conventional laparoscopic approach as therapy for uterovaginal prolapse. Surgical techniques, efficacy and overall results are compared.

Methods:

In this prospective study 40 consecutive patients with uro-genital prolapse are randomized to sacropexy: 20 by an open approach, 20 by a conventional laparoscopy approach. Anchorage is achieved in both groups by two polypropylene meshes.

Check-ups were scheduled at 3, 6, 12 months and then yearly. Pre-operative patient characteristics, operative and post-operative events and follow-up results are recorded.

DETAILED DESCRIPTION:
Surgical technique In both open or laparoscopic approach the anterior vaginal wall is dissected from the bladder to expose a vaginal wall area of at least 3 x 5 cms where the mesh will be attached with four-five Polyglycolic 0 sutures. The procedure is repeated for the posterior vaginal wall, where the mesh will be attached with three-four Polyglycolic 0 sutures.

The sacral promontory surface is prepared and 1 or 2 non-reabsorbable 0.0 sutures are placed into the sacral periosteum about 2 cm below the promontory. A sub-peritoneal tunnel is created through which meshes are passed avoiding traction to the sacrum. The peritoneum is closed over the meshes.

ELIGIBILITY:
Inclusion Criteria:

* Study inclusion criteria were POP > 2, age ≥ 18 and ≤ 75 yrs.

Exclusion Criteria:

* Malignant uterus lesion (leiomyoma, fibromyoma, cervical or endometrial carcinoma)

  * Active pelvic inflammatory disease,
  * Known hypersensitivity to synthetic materials (polypropylene or polyglycolic acid)
  * Pregnancy or lactation
  * Evidence of clinically significant cardiovascular, renal, hepatic or respiratory diseases; and
  * Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Operative morbidity and adverse events | 2 years
  Operative morbidity according to Clavien-Dindo classification, measure of perioperative pain with Visual Analogue Score VAS, post-operative adverse events constitute the outcome measures, together with operating time, intra-operative blood loss and length of hospital stay.

SECONDARY OUTCOMES:
Subjective and objective success rate, Patient satisfaction | 2 years
  Success rate: subjective success is absence of symptoms related to prolapse or incontinence using Urogenital Distress Inventory (URI-6) and Impact Incontinence Quality of Life (IIQ-7). Patient satisfaction is defined by replies to the questions of whether the patient is satisfied and would repeat the operation. Objective success is defined as no vaginal prolapse greater or equal to grade 2 at any vaginal site, while the patient performed Valsalva's manouever.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Porena, MD Prof in Chief, Study Director — Department of Medical-Surgical Specialties and Public Health, Section of Urology and Andrology
Locations (1):
- Department of Medical-Surgical Specialties and Public Health, Section of Urology and Andrology, Perugia, Italy

REFERENCES:
- [Background] Costantini E, Mearini L, Bini V, Zucchi A, Mearini E, Porena M. Uterus preservation in surgical correction of urogenital prolapse. Eur Urol. 2005 Oct;48(4):642-9. doi: 10.1016/j.eururo.2005.04.022. PMID 15964131
- [Background] Costantini E, Zucchi A, Giannantoni A, Mearini L, Bini V, Porena M. Must colposuspension be associated with sacropexy to prevent postoperative urinary incontinence? Eur Urol. 2007 Mar;51(3):788-94. doi: 10.1016/j.eururo.2006.08.034. Epub 2006 Sep 5. PMID 17011699
- [Background] Costantini E, Lazzeri M, Bini V, Del Zingaro M, Zucchi A, Porena M. Burch colposuspension does not provide any additional benefit to pelvic organ prolapse repair in patients with urinary incontinence: a randomized surgical trial. J Urol. 2008 Sep;180(3):1007-12. doi: 10.1016/j.juro.2008.05.023. Epub 2008 Jul 17. PMID 18639302
- See also: university of perugia — http://www.unipg.it